CLINICAL TRIAL: NCT04294992
Title: Granisteron Versus Ondansetron for Prophylaxis Against Post-Spinal Anesthesia Shivering: a Randomized Controlled Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Ayman Abougabal, lecturer of anaesthesia, SICU and pain management, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MS-265-2019
Record Dates: First submitted 2020-03-02; First posted 2020-03-04 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Spinal Anaesthetic
MeSH Terms: interventions — Ondansetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Granisteron group (Experimental)
  Interventions: Drug: Ondansetron 8mg
- Ondansetron group (Active Comparator)
  Interventions: Drug: Ondansetron 8mg

INTERVENTIONS:
Drug: Ondansetron 8mg — Study drugs will be prepared, diluted to a volume of 10 mL using saline 0.9%

SUMMARY:
3. Scientific committee approval (Was it scientifically approved by the department?) Yes

Date of approval: Sunday ,1ST September,2019

Background and Rationale:

Regional anesthesia is commonly associated with intraoperative shivering which reaches 40-60%. Spinal anesthesia contributes in impairment of thermoregulation, and predisposes patients to hypothermia, which reduces the threshold for shivering and vasoconstriction. Other mechanisms responsible for shivering include increased sympathetic tone, pain, and systemic release of pyrogens. Shivering causes increase in metabolic activity, oxygen consumption, intracranial, and intraocular pressure. Shivering is also responsible for increasing cardiac output, peripheral resistance, carbon dioxide production, and lactic acidosis. Furthermore, shivering interferes with electrocardiogram (ECG) and pulse oximetry. 1 Post anaesthetic shivering is one of the most frequent problems in the early recovery phase following general anaesthesia. It was considered as the sixth most important problem of current clinical anaesthesiology among 33 low morbidity clinical outcomes. Previous studies have found that shivering occurs up to 60% of patients in the postoperative period and varies according to sex, age, drugs used for anaesthesia and the duration for the surgery.2 Since shivering is a response to hypothermia, body temperature should be maintained within 36.5-37.5°C, however, shivering may be also seen in normothermic patients undergoing regional anesthesia. A number of factors responsible for developing of hypothermia in regional anesthesia including age, level of sensory block, temperature of the operating room and infusion solution.3 Perioperative hypothermia and shivering can be prevented by physical methods like surface warming or pharmacologically by drugs such as pethidine, tramadol, clonidine, doxapram, opioids, neostigmine, magnesium sulfate and ketamine.4 Pethidine is the most commonly used drug for post spinal anesthesia shivering. The disadvantage of pethidine is that it can cause respiratory depression in the presence of previously administered opioids or anaesthetics. Moreover, hypotension, nausea and vomiting are also important side effect of pethidine.5 Pethidine, which is considered as a time-tested drug for control of shivering, can have adverse effects such as respiratory depression, nausea, and vomiting. which begs to investigate the efficacy of other drugs.6 5-HT antagonists had been effectively introduced for management of perioperative shivering by inhibiting thermoregulatory response by central mechanism. Ondansetron is a 5-HT antagonist which had been effectively used in treatment of postoperative shivering.7 Granisteron, a new generation of 5-HT antagonists, had been also reported effective in the prevention of Postoperative shivering.9-10 No data are available about the comparison of both drugs, ondansetron and granisteron, for prophylaxis against post-spinal shivering The aim of the investigator's study is to compare the efficacy of granisteron to ondansetron for prevention of intra- and post spinal anaesthesia shivering.

ELIGIBILITY:
Inclusion Criteria:

* • With ASA physical status I and II

  * Scheduled to undergo lower half surgery under spinal anesthesia such as lower limb orthopedic surgeries, lower limb plastic surgeries, or lower abdominal surgeries.

Exclusion Criteria:

* • Patient refusal

  * Patients with age above 60 years and below 18 years.
  * Pregnant
  * Patients with contraindications to spinal anesthesia
  * Preoperative fever or hypothermia (temperature >38°C or below 36.5°C), hypo or hyperthyroidism, a requirement for blood or blood product transfusion during surgery and medications likely to alter thermoregulation or nausea and vomiting, will be excluded.
  * Patients with significant cardiopulmonary disease (i.e. ejection fraction <40% and/or SpO2 < 92% on room air) or psychological disorder
  * impaired renal (serum creatinine > 2 mg/dL) or hepatic function (class B or C on Child-Pugh score)
  * Procedures with anticipated duration less than 90 minutes or more than 180 min, those received saddle block or those required vasodilator administration
  * Allergy to any of the study drugs will be excluded from the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
perioperative spinal induced shivering | during spinal anaesthesia
  incidence of shivering during spinal anaesthsia

SECONDARY OUTCOMES:
incidence of perioperative nausea and vomiting | during spinal anaethesia

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nallam SR, Cherukuru K, Sateesh G. Efficacy of Intravenous Ondansetron for Prevention of Postspinal Shivering during Lower Segment Cesarean Section: A Double-Blinded Randomized Trial. Anesth Essays Res. 2017 Apr-Jun;11(2):508-513. doi: 10.4103/aer.AER_26_17. PMID 28663651
- [Background] Iqbal A, Ahmed A, Rudra A, Wankhede RG, Sengupta S, Das T, Roy D. Prophylactic granisetron vs pethidine for the prevention of postoperative shivering: a randomized control trial. Indian J Anaesth. 2009 Jun;53(3):330-4. PMID 20640142